CLINICAL TRIAL: NCT06073431
Title: Longitudinal Observational Trial to Uncover Subtypes of Cancer Cachexia
Brief Title: LOTUS-CC: An Observational Research Study to Uncover Subtypes of Cancer Cachexia
Acronym: LOTUS
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Dunne, URCC Study Chair, University of Rochester
Other Study IDs: URCC-22063; NCI-2023-04268 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC-22063 (Other: University of Rochester NCORP Research Base); URCC-22063 (Other: DCP); URCC-22063 (Other: CTEP); UG1CA189961 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Advanced Colorectal Carcinoma; Advanced Lung Non-Small Cell Carcinoma; Advanced Pancreatic Adenocarcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Colorectal Carcinoma; Unresectable Lung Non-Small Cell Carcinoma; Unresectable Pancreatic Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms | interventions — Specimen Handling; Exercise Test; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey, function tests, biospecimen, actigraph): Patients complete surveys over 30 minutes, undergo physical function tests over 30 minutes, undergo collection of blood and archived tumor samples, and wear actigraph over 24 hours for 7 days to record daily sleep and exercise activity at baseline and 3-month follow-up. Additionally, patients undergo standard of care CT or PET/CT scans throughout the study and patients' medical records are also reviewed at baseline, 3-month and 1-year follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Procedure: Positron Emission Tomography; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and archived tumor samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Electronic Health Record Review — Medical records reviewed
Other: Medical Device Usage and Evaluation — Wear actigraph
Other: Physical Performance Testing — Undergo physical function tests
  Other Names: Physical Fitness Testing; Physical Function Testing
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates cancer-related weight and muscle mass loss, symptoms, and physical function (cachexia) in patients undergoing treatment for colorectal, lung, or pancreatic cancer that cannot be removed by surgery (unresectable) or is stage IV. Patients with these cancer types are at risk for developing cancer cachexia (CC), which is defined as weight loss, muscle loss, and fat loss due to cancer. CC has been associated with reduced physical performance, impaired quality of life, and poorer survival. Many studies that have evaluated treatments for cancer-related weight and muscle loss have aimed to treat all patients with weight loss exactly the same and, unfortunately, have not been successful. Like different cancer types, weight and muscle loss related to cancer may have different causes in different individuals and the best treatment strategy for this condition may not be a one-size-fits-all approach. Information gathered from this study may help researchers develop new diagnostic criteria for CC and design better treatments and clinical trials for cancer-related weight and muscle loss in the future to improve the quality of life in patients with advanced colorectal, lung, or pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify multiple distinct diagnostic subtypes within the syndrome of CC as defined by host characteristics (e.g. cachexia symptoms, physical activity, physical function, blood biomarkers including hemoglobin and albumin, and body composition) at baseline and change in these factors over time in patients with cancer at high risk for CC.

SECONDARY OBJECTIVES:

I. To determine the association of each CC phenotype with overall survival. II. To validate CC diagnostic phenotypes developed in a separate, independent cachexia observational study performed by our collaborators at Kaiser Permanente.

III. To collect human samples of blood, tumor tissue, and medical images and build a large, comprehensive CC database clinically annotated with cancer-related outcomes, cachexia symptoms, and physical function data.

EXPLORATORY OBJECTIVE:

I. To evaluate for tumor-derived factors contributing to CC by determining the association between interleukin-6 (IL-6) expression in tumor and IL-6 and CC chemokine ligand 2 (CCL2) levels in the blood in patients with CC.

OUTLINE: This is an observational study.

Patients complete surveys over 30 minutes, undergo physical function tests over 30 minutes, undergo collection of blood and archived tumor samples, and wear actigraph over 24 hours for 7 days to record daily sleep and exercise activity at baseline and 3-month follow-up. Additionally, patients undergo standard of care computed tomography (CT) or positron emission tomography (PET)/CT scans throughout the study and patients' medical records are also reviewed at baseline, 3-month and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of unresectable or stage IV 1) non-small cell lung cancer (NSCLC), 2) pancreatic adenocarcinoma, or 3) colorectal cancer

  * Note: Patients do not need to have cachexia to be eligible
* Plan to start first-line systemic anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, interventional clinical trial) in the next 6 weeks or has started first-line systemic therapy in the previous 6 weeks.

  * NOTE: Patients who received systemic anti-cancer therapy previously as part of adjuvant or neoadjuvant treatment and have since recurred are still eligible if such treatment ended > 6 months prior to enrollment. Patients receiving concurrent radiation with systemic therapy or received local therapy alone (surgery, radiation therapy [RT]) prior to first line therapy remain eligible. Patients receiving maintenance treatment after first line therapy are not eligible
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Be able to understand, speak and read English
* Be 18 years of age or older

Exclusion Criteria:

* Have contraindications to physical function assessments (30-second arm curl, Timed-Up-And-Go test, or 30-second chair-stand test) per the treating provider or their designee
* Have any planned major surgeries within the next 3 months
* Have received chemotherapy or surgery for separate primary cancer within the past 3 years other than early local staged non-melanoma skin cancer
* Be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment for non-small cell lung cancer (NSCLC), pancreatic adenocarcinoma, colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-11-13 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of multiple distinct diagnostic subtypes within the syndrome of cancer cachexia (CC) | Baseline through study completion, assessed up to 1 year follow up
  Defined by host characteristics (e.g. cachexia symptoms, physical activity, physical function, blood biomarkers including hemoglobin and albumin, and body composition) at baseline and change in these factors over time in patients with cancer at high risk for CC. First, will examine the distributions of each variable and assess the need for using transformations to achieve normality for continuous variables (log transformation, quartiles, or clinically important thresholds), collapsing similar variables into single categories, and excluding conditions that are too rare (< 1% of the cohort). Next, will assess statistical correlations using the Jaccard similarity metric for binary variables and the Pearson or Spearman correlation for continuous variables to determine highly correlated variables that may provide redundant information.

SECONDARY OUTCOMES:
Association of each CC phenotype (clusters) with overall survival | Days from registration (day 0) to death (the event) or the last contact (censored), assessed up to 1 year follow up
  Will be assessed in the Cox regression model. Will estimate the bivariate association where the only independent variables will be the indicators for the cluster membership. Will report the hazard ratio for the association of each CC phenotype, specifying the lowest-risk cluster as the reference. Will assess the influence of selected factors (e.g., age, performance status, and other known prognostic factors) on the association of the cluster with survival by adding the factor to the model as a covariate and keeping those that resulted in 10% or more change in any regression coefficients for cluster membership. Will assess if the association of clusters with survival varies by specific subgroups (e.g., older versus younger age, gender, and cancer type). Will assess the statistical significance interaction of the subgroup with the cluster membership by maximum likelihood test and evaluate the regression coefficients for clusters in each subgroup comparing the direction and magnitude.
Validation of CC diagnostic phenotypes developed in a separate, independent cachexia observational study performed by collaborators at Kaiser Permanente | Up to study completion, assessed up to 1 year
  Study participants will be categorized into the Kaiser Permanente Northern California (KPNC)-derived CC phenotype groups. Will use the final latent class analysis model fit in the KPNC data to compute the posterior probabilities of membership in each latent class for each individual National Cancer Institute Community Oncology Research Program (NCORP) participant based on his/her individual data. Will compare cluster prevalence in each cohort as well as the distributions of the variables used to determine each cluster to investigate patterns of commonality and dissimilarity across the contributing variables. Validation will be determined by fitting University of Rochester Cancer Center (URCC) NCORP participants in KPNC-derived clusters and evaluating each cluster's association with survival. If the ranking of survival (best to worst) among each cluster in the URCC NCORP dataset mirrors the prognostic ranking of clusters in the KPNC dataset, the clusters will be deemed validated.

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Dunne, Principal Investigator — University of Rochester NCORP Research Base
Locations (225):
- United States (225):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - The Longstreet Clinic - Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Tift Regional Medical Center, Tifton, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Health Center - Greenfield, Greenfield, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin